CLINICAL TRIAL: NCT00311883
Title: Phase 1 Study of Hydroxychloroquine in Cystic Fibrosis
Brief Title: Hydroxychloroquine in Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Bonnie Slovis, M.D., Vanderbilt University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060051
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Induced sputum; Lung inflammation
MeSH Terms: conditions — Cystic Fibrosis; Pneumonia | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: hydroxychloroquine

SUMMARY:
Study levels of inflammatory mediators in induced sputum of patients with cystic fibrosis before and after a 4 week course of oral hydroxychloroquine.

DETAILED DESCRIPTION:
Open label study of effect of hydroxychloroquine on inflammation, bacterial burden and exhaled breath condensate pH in patients with cystic fibrosis. Patients with cystic fibrosis, 16 years or older and with pulmonary function tests with an FEV1 greater than 40% predicted will be eligible for enrollment. Enrolled subjects will undergo collection of exhaled breath condensate and sputum induction and collection following nebulized hypertonic saline, before and following a 4 week course of oral hydroxychloroquine at 200 mg a day. Inflammatory mediators, neutrophil counts, and bacterial density in sputum and exhaled breath condensate pH will be measure at entry and at the end of 4 weeks of oral drug. There will be no placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 16 years and 65 years of age.
2. Confirmed diagnosis of CF based on the following criteria:

   i. positive sweat chloride 60 mEq/liter (by pilocarpine iontophoresis) and/or ii. a genotype with two identifiable mutations consistent with CF, and iii. accompanied by one or more clinical features consistent with the CF phenotype
3. FEV1 50% predicted value (subjects 16- <18 years of age) or 40% predicted value (subjects 18 years of age)
4. Clinically stable with no evidence of acute upper or lower respiratory tract infection or current pulmonary exacerbation within the 14 days prior to Visit 1 (Day 0)
5. Ability to reproducibly perform spirometry and peak flow measurements
6. Ability to understand and sign a written informed consent or assent and comply with the requirements of the study

Exclusion Criteria:

1. Use of an investigational agent within the 4-week period prior to Visit 1
2. Chronic daily use of ibuprofen or other NSAIDs, or systemic corticosteroids, or any oral diabetic or hypoglycemic agent within the 4 weeks prior to Visit 1 or acute usage within 72 hours prior to Visit 1
3. History of hypersensitivity to beta-agonists
4. History of hypersensitivity to hydroxychloroquine or chloroquine
5. Oxygen saturation < 92% on room air at Visit 1
6. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
7. History of hemoptysis 30 cc per episode during the 30 days prior to Visit 1
8. Significant history of hepatic, cardiovascular, renal, neurological, hematologic, or peptic ulcer disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory mediators and exhaled breath condensate pH following 4 week administration of drug. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie S Slovis, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States